CLINICAL TRIAL: NCT05071599
Title: Assessment of the Efficacy of Twin Arch Brackets in the Control of Orthodontic Tooth Movement: A Randomized Controlled Clinical Study
Brief Title: Efficacy of Twin Arch Brackets in the Control of Orthodontic Tooth Movement
Acronym: TAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohammed Basher Farhat, Dentist, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Twin arch brackets
Record Dates: First submitted 2021-09-12; First posted 2021-10-08 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Orthodontic Tooth Movement
Keywords: Brackets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin arch brackets (Experimental): the malocclusion for this group will be treated using fixed appliance which utilize twin arch brackets system.
  Interventions: Device: Twin Arch Brackets
- Conventional brackets (Experimental): the malocclusion for this group will be treated using fixed appliance which utilize conventional "pre-adjusted edgewise "brackets system.
  Interventions: Device: Twin Arch Brackets

INTERVENTIONS:
Device: Twin Arch Brackets — Twin Arch Brackets characterized by double horizontal slots which make it capable to accept two arch wire at the same time which in turn can achieve a better control over orthodontic tooth movement
  Other Names: Preadjusted Edgewise Brackets

SUMMARY:
To evaluate the efficacy of twin arch brackets compared to conventional brackets in the control of orthodontic tooth movement.

DETAILED DESCRIPTION:
Alignment and leveling of teeth generally constitute the most important preliminary clinical phase of any orthodontic treatment with fixed orthodontic appliances.

During the leveling and alignment stage, tooth movement is directly affected by many factors, such as interbracket distance, bracket width, archwire selection and the friction generated between the bracket and the archwire. It is critical that the force moment which generated by interaction between the bracket slot and the archwire to be transferred from the archwire to the malpositioned tooth.

While it is widely recognized that the geometric structure of the bracket, especially the slot width, determines the efficiency of the force moment, the interbracket span, on the other hand, remains another crucial factor affecting the effectiveness of tooth displacement. It has been established that a sufficient interbracket span enables the flexible archwire to activate its springiness caused by deflection. A wider bracket is favorable to develop an adequate force moment, but the subsequent decrease in the space between the brackets will reduce the effective length of the archwire segments between the supports. As a matter of fact, the efficiency of treatment mechanics is a major focus in modern orthodontics.The advancement of bracket design began with the vertically positioned slot in the ribbon arch appliance to the pure rectangular horizontal slot in the traditional standard edgewise to the modern preadjusted brackets in the straight wire technique, and to the current design of the self-ligating brackets system. It is interesting to note that despite the numerous bracket designs, one feature has remained unchanged: there is only one single horizontal slot on the facial surface of the bracket. In some design variations, such as the Tip- Edge Plus, In-Ovation and " R " brackets, an additional horizontal slot is enclosed within the bracket base and is not open to the labial surface, therefore only allowing for engagement of segmental auxiliary archwires. However some inventors design bracket system called "the twin wire appliance or twin arch wire appliance " which can fit two archwires simultaneously by incorporating two horizontal slots in the design of single brackets. In twin arch appliance design, the bracket width is doubled without decreasing the interbracket span.

The treatment technique to work with two arch wires simultaneously is not new. The idea behind the invention of twin arch appliance was to achieve a better control over orthodontics tooth movements. In the orthodontic literature a very little knowledge and research can be found concerning the use of Twin arch appliance in orthodontic treatment. In the 1930s attempts were made to develop a new treatment method with this concept. Spencer Atkinson was the pioneer, Spencer created a bracket with a vertical and a horizontal slot, positioned one on top of the other. Then in 2008 an experimental study for the efficiency of double slot brackets in correction of malposed teeth when placed in wax typodont was established. The study revealed that twin slot bracket doubles the rate of teeth alignment. The reason behind this phenomenon that the twin-slot bracket doubles the rate of alignment may be attributed to fact that the force applied on the tooth bonded with the twin-slot bracket is doubled and the rate of wax flow is likely to be proportional to load .

Because of the promising results obtained from the previous experimental study and the lack of clinical study results, it will be beneficial to study and compare clinically the effectiveness of twin arch appliance in control of orthodontic tooth movements as well as the comfort of patient during the initial leveling and alignment stage of treatment in relation to other conventional bracket systems.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 13 to 18 years.
2. Full set of permanent teeth (the third molars are not considered).
3. Angle class I malocclusion with normal facial proportions.
4. Mild to moderate crowding in both arches that require treatment with fixed appliance using non extraction approach
5. No previous orthodontic or orthognathic surgery treatment.
6. Free from oral and general health problems that could interfere with orthodontic treatment..
7. All teeth should be caries-free.

Exclusion Criteria:

1. Patients with poor oral hygiene or periodontally compromised teeth.
2. History of serious medical problems or taking systemic medication which could affect orthodontic treatment.
3. History of serious dental problems (endodontic treatment, periodontal surgery, apicectomy, or any other dental problems) which could affect orthodontic treatment.
4. History of trauma, bruxism, or or parafunctional habits.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy of Twin Arch brackets in orthodontic tooth movement | 1 years
  Time taken for leveling and alignment phase for anterior teeth will be evaluated for each group.

SECONDARY OUTCOMES:
Comfort of Twin Arch brackets . | 1 week
  Pain in day 1 to day 7 after brackets and archwires placement will be evaluated for each group of patients.
Patient acceptance or preference. | 1 year
  Patient acceptance or preference for the sight of brackets will be evaluated for each group
Failure of brackets bonding | 2 years
  Number of brackets debonding or fracture during treatment period will be evaluated and recorded monthly for each group of patients
Oral hygiene maintenance | 1.5 year
  Patient capability to keep up with oral hygiene measures and instructions will be evaluated for each group of patients

CONTACTS AND LOCATIONS:
Overall Officials: Raafat E G Mohamed, Asst Prof, Study Director — Department of orthodontics, Faculty of Dental Medicine (Boys-Cairo), Al-Azhar University; Ahmed S Ammar, Lecturer, Study Director — Department of Orthodontics, Faculty of Dental Medicine (Boys- Cairo), Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
When the research done and I finished my master degree the research will available for the public
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 - 3 years
Access Criteria: Via email massages

REFERENCES:
- [Background] Gravina MA, Brunharo IH, Fraga MR, Artese F, Campos MJ, Vitral RW, Quintao CC. Clinical evaluation of dental alignment and leveling with three different types of orthodontic wires. Dental Press J Orthod. 2013 Nov-Dec;18(6):31-7. doi: 10.1590/s2176-94512013000600006. PMID 24351147
- [Background] Sifakakis I, Pandis N, Makou M, Eliades T, Katsaros C, Bourauel C. A comparative assessment of torque generated by lingual and conventional brackets. Eur J Orthod. 2013 Jun;35(3):375-80. doi: 10.1093/ejo/cjs029. Epub 2012 May 9. PMID 22573909
- [Background] Khattab TZ, Hajeer MY, Farah H, Al-Sabbagh R. Maxillary dental arch changes following the leveling and alignment stage with lingual and labial orthodontic appliances: a preliminary report of a randomized controlled trial. J Contemp Dent Pract. 2014 Sep 1;15(5):561-6. doi: 10.5005/jp-journals-10024-1579. PMID 25707826
- [Background] Liaw YC, Su YY, Lai YL, Lee SY. Stiffness and frictional resistance of a superelastic nickel-titanium orthodontic wire with low-stress hysteresis. Am J Orthod Dentofacial Orthop. 2007 May;131(5):578.e12-8. doi: 10.1016/j.ajodo.2006.08.015. PMID 17482074
- [Background] Shen G, Chen RJ, Hu Z, Qian YF. The effects of a newly designed twin-slot bracket on severely malpositioned teeth--a typodont experimental study. Eur J Orthod. 2008 Aug;30(4):401-6. doi: 10.1093/ejo/cjn011. PMID 18678759
- [Background] Miles PG, Weyant RJ, Rustveld L. A clinical trial of Damon 2 vs conventional twin brackets during initial alignment. Angle Orthod. 2006 May;76(3):480-5. doi: 10.1043/0003-3219(2006)076[0480:ACTODV]2.0.CO;2. PMID 16637731
- [Background] Yeh CL, Kusnoto B, Viana G, Evans CA, Drummond JL. In-vitro evaluation of frictional resistance between brackets with passive-ligation designs. Am J Orthod Dentofacial Orthop. 2007 Jun;131(6):704.e11-22. doi: 10.1016/j.ajodo.2006.09.041. PMID 17561042
- [Background] Rinchuse DJ, Rinchuse DJ, Kapur-Wadhwa R. Orthodontic appliance design. Am J Orthod Dentofacial Orthop. 2007 Jan;131(1):76-82. doi: 10.1016/j.ajodo.2005.04.039. No abstract available. PMID 17208110
- [Background] Parkhouse RC. Current products and practice: Tip-Edge Plus. J Orthod. 2007 Mar;34(1):59-68. doi: 10.1179/146531207225021933. PMID 17347298
- [Background] Miles P, Weyant R. Porcelain brackets during initial alignment: are self-ligating cosmetic brackets more efficient? Aust Orthod J. 2010 May;26(1):21-6. PMID 20575195
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- See also: Clinical evaluation of the failure rates of metallic brackets — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3894768/
- See also: A COMPARISON STUDY OF BRACKET FAILURE RATE BETWEEN DIRECT AND INDIRECT BONDING TECHNIQUES — https://ajdsm.journals.ekb.eg/article_108468_7c1e0df081158d3f51a0f82c688d143c.pdf